CLINICAL TRIAL: NCT04367259
Title: Comparison of the Efficacy of Single and Double Puncture Arthrocentesis in Treatment of Temporomandibular Joint Disc Displacement Without Reduction
Brief Title: Single Puncture Arthrocentesis vs Double Puncture Arthrocentesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, Fatih TASKESEN, Head of Dept. Oral and Maxillofacial Surgery, Erzincan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 135163
Record Dates: First submitted 2020-04-03; First posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Arthrocentesis
Keywords: Temporomandibular Joint
MeSH Terms: interventions — Arthrocentesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single puncture arthrocentesis (SPA) group (Active Comparator): Patients presenting temporomandibular joint disc displacement without reduction (DDwoR) treated with single puncture arthrocentesis
  Interventions: Procedure: TMJ Arthrocentesis
- Double puncture arthrocentesis (DPA) group (Active Comparator): Patients presenting temporomandibular joint disc displacement without reduction (DDwoR) treated with double puncture arthrocentesis
  Interventions: Procedure: TMJ Arthrocentesis

INTERVENTIONS:
Procedure: TMJ Arthrocentesis — Temporomandibular joint arthrocentesis

SUMMARY:
The aim of the present study was to compare the treatment efficacy of single puncture arthrocentesis (SPA) and double puncture arthrocentesis (DPA) techniques in Temporomandibular joint (TMJ) disc displacement without reduction (DDwoR).

DETAILED DESCRIPTION:
Study sample consisted of 36 patients with DDwoR. 18 patients received SPA procedure and included in SPA group. The other 18 patients received DPA procedure and included in DPA group.

Double puncture arthrocentesis technique:

Posterior puncture method was used as described by Alkan and Etoz. for DPA. A straight line was drawn with a marker pen along the skin from the middle portion of the auricular tragus to the lateral chantus. The first puncture point was marked 10 mm anterior and 2 mm inferior to the tragus and the second 7 mm anterior and 2 mm inferior to the tragus. After local anesthesia, upper joint cavity was irrigated with 200 mL of Lactated Ringer's (RL) solution by inserting two 21- gauge needle. At the end of the procedure, after withdrawn of one of the needles, 1 mL of sodium hyaluronate (SH) was injected into the upper TMJ compartment through the other needle.

Single Puncture Arthrocentesis Technique:

SPA was performed with one needle (SPA Type-1 according to Senturk and Cambazoglu). The first reference point in DPA was used as the needle entry point fort he SPA. With this technique, the inflow and outflow of solution were provided through the same cannula and lumen of one 21-gauge needle as described by Guarda-Nardini et al. The joint was irrigated with 200 mL of RL solution under high pressure. At the end of the procedure1 mL of SH was injected through the needle.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Temporomandibular joint (TMJ) disc displacement without reduction.
* Restricted mouth opening

Exclusion criteria:

* History of systemic disease effecting TMJ.
* History of previous TMJ surgery

Ages: 21 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
The Rate of Pain on Function (PoF) assessed by Numerical Rating Scale (NRS) | baseline (t0)
  Patients rated their pain on function (pain during chewing or speaking etc.) on a Numeric Rating Scale (NRS) (0-10 where 0 is no pain and 10 is the worst pain imaginable)
The Rate of Pain on Function (PoF) assessed by Numerical Rating Scale (NRS) | At 1st week (t1)
  Patients rated their pain on function (pain during chewing or speaking etc.) on a Numeric Rating Scale (NRS) (0-10 where 0 is no pain and 10 is the worst pain imaginable)
The Rate of Pain on Function (PoF) assessed by Numerical Rating Scale (NRS) | at 1st month (t2)
  Patients rated their pain on function (pain during chewing or speaking etc.) on a Numeric Rating Scale (NRS) (0-10 where 0 is no pain and 10 is the worst pain imaginable)
The Rate of Pain on Function (PoF) assessed by Numerical Rating Scale (NRS) | at 3rd month (t3)
  Patients rated their pain on function (pain during chewing or speaking etc.) on a Numeric Rating Scale (NRS) (0-10 where 0 is no pain and 10 is the worst pain imaginable)
The Rate of Pain on Function (PoF) assessed by Numerical Rating Scale (NRS) | at 6th month (t4)
  Patients rated their pain on function (pain during chewing or speaking etc.) on a Numeric Rating Scale (NRS) (0-10 where 0 is no pain and 10 is the worst pain imaginable)
The measurement of pain-free maximum mouth opening (MMO) in millimeters | baseline (t0)
  Pain-free MMO was measured as the distance between the incisal edges of the upper and lower incisors while patient's mouth is open as possible without any assistance and without pain. Three measurements were performed, and their average is recorded.
The measurement of pain-free maximum mouth opening (MMO) in millimeters | at 1st week (t1)
  Pain-free MMO was measured as the distance between the incisal edges of the upper and lower incisors while patient's mouth is open as possible without any assistance and without pain. Three measurements were performed, and their average is recorded.
The measurement of pain-free maximum mouth opening (MMO) in millimeters | at 1st month (t2)
  Pain-free MMO was measured as the distance between the incisal edges of the upper and lower incisors while patient's mouth is open as possible without any assistance and without pain. Three measurements were performed, and their average is recorded.
The measurement of pain-free maximum mouth opening (MMO) in millimeters | at 3rd month (t3)
  Pain-free MMO was measured as the distance between the incisal edges of the upper and lower incisors while patient's mouth is open as possible without any assistance and without pain. Three measurements were performed, and their average is recorded.
The measurement of pain-free maximum mouth opening (MMO) in millimeters | at 6th month (t4)
  Pain-free MMO was measured as the distance between the incisal edges of the upper and lower incisors while patient's mouth is open as possible without any assistance and without pain. Three measurements were performed, and their average is recorded.

SECONDARY OUTCOMES:
The rate of pain at rest (PaR) assessed by Numerical Rating Scale (NRS) | At Baseline (t0)
  Patients rated their pain level at rest on a Numerical pain Scale (NRS) )(0-10 where 0 is no pain and 10 is the worst pain imaginable)
The rate of pain at rest (PaR) assessed by Numerical Rating Scale (NRS) | at 1st week (t1)
  Patients rated their pain level at rest on a Numerical pain Scale (NRS) )(0-10 where 0 is no pain and 10 is the worst pain imaginable)
The rate of pain at rest (PaR) assessed by Numerical Rating Scale (NRS) | at 1st month (t2)
  Patients rated their pain level at rest on a Numerical pain Scale (NRS) )(0-10 where 0 is no pain and 10 is the worst pain imaginable)
The rate of pain at rest (PaR) assessed by Numerical Rating Scale (NRS) | at 3rd month (t3)
  Patients rated their pain level at rest on a Numerical pain Scale (NRS) )(0-10 where 0 is no pain and 10 is the worst pain imaginable)
The rate of pain at rest (PaR) assessed by Numerical Rating Scale (NRS) | at 6th month (t4)
  Patients rated their pain level at rest on a Numerical pain Scale (NRS) )(0-10 where 0 is no pain and 10 is the worst pain imaginable)
Measurement of Duration of the Procedure in Minutes | at 1st day (At the end of the procedure)
  Total time for arthrocentesis was noted at the end of the procedure
Measurement of the easiness of the procedure to the operator by using Visual Analog Scale (VAS) | at 1st day (At the end of the procedure)
  The operator rated the degree of easiness of the procedure on a VAS as 0-very easy 10-very difficult to perform.
The rate of treatment tolerability assessed by 5-point Likert-type scale | 1st day
  The degree to which overt adverse effects and post operative complications (pain, feeling of pressure in TMJ area and disturbing sound) can be tolerated by the patient. Patients were asked to rate the tolerability on a 5 point scale as 0- lowest, 4-highest.
The rate of treatment tolerability assessed by 5-point Likert-type scale | 1st week
  The degree to which overt adverse effects and post operative complications (pain, feeling of pressure in TMJ area and disturbing sound) can be tolerated by the patient. Patients were asked to rate the tolerability on a 5 point scale as 0- lowest, 4-highest.
The rate of treatment tolerability assessed by 5-point Likert-type scale | 6th month
  The degree to which overt adverse effects and post operative complications (pain, feeling of pressure in TMJ area and disturbing sound) can be tolerated by the patient. Patients were asked to rate the tolerability on a 5 point scale as 0- lowest, 4-highest.
The rate of chewing efficiency by using Visual Analog Scale (VAS) | at baseline (t0)
  Patients rated the chewing efficiency on a VAS as 0-can only eat semi-liquid foods, 10-eat any solid-food.
The rate of chewing efficiency by using Visual Analog Scale (VAS) | at 1st week (t1)
  Patients rated the chewing efficiency on a VAS as 0-can only eat semi-liquid foods, 10-eat any solid-food.
The rate of chewing efficiency by using Visual Analog Scale (VAS) | at 1st month (t2)
  Patients rated the chewing efficiency on a VAS as 0-can only eat semi-liquid foods, 10-eat any solid-food.
The rate of chewing efficiency by using Visual Analog Scale (VAS) | at 3rd month (t3)
  Patients rated the chewing efficiency on a VAS as 0-can only eat semi-liquid foods, 10-eat any solid-food.
The rate of chewing efficiency by using Visual Analog Scale (VAS) | at 6th month (t4)
  Patients rated the chewing efficiency on a VAS as 0-can only eat semi-liquid foods, 10-eat any solid-food.
Rate of perceived effectiveness of the treatment by using 5-point Likert-type scale | at 6th month
  Patients rated the subjective treatment effectiveness on a 5-point scale as 0- lowest, 4 highest values.
Measurement of Lateral Movement of the mandible towards the affected Temporomandibular joint (TMJ) in millimeters | at baseline (t0)
  Lateral Movement of the mandible towards the affected Temporomandibular joint (LT) was measured as the distance between the midlines of the upper and lower incisors by a caliper while patient's mandible was shifted towards the affected TMJ. Three measurements were performed, and their average is recorded.
Measurement of Lateral Movement of the mandible towards the affected Temporomandibular joint (TMJ) in millimeters | at 1st week (t1)
  Lateral Movement of the mandible towards the affected Temporomandibular joint (LT) was measured as the distance between the midlines of the upper and lower incisors by a caliper while patient's mandible was shifted towards the affected TMJ. Three measurements were performed, and their average is recorded.
Measurement of Lateral Movement of the mandible towards the affected Temporomandibular joint (TMJ) in millimeters | at 1st month (t2)
  Lateral Movement of the mandible towards the affected Temporomandibular joint (LT) was measured as the distance between the midlines of the upper and lower incisors by a caliper while patient's mandible was shifted towards the affected TMJ. Three measurements were performed, and their average is recorded.
Measurement of Lateral Movement of the mandible towards the affected Temporomandibular joint (TMJ) in millimeters | at 3rd month (t3)
  Lateral Movement of the mandible towards the affected Temporomandibular joint (LT) was measured as the distance between the midlines of the upper and lower incisors by a caliper while patient's mandible was shifted towards the affected TMJ. Three measurements were performed, and their average is recorded.
Measurement of Lateral Movement of the mandible towards the affected Temporomandibular joint (TMJ) in millimeters | at 6th month (t4)
  Lateral Movement of the mandible towards the affected Temporomandibular joint (LT) was measured as the distance between the midlines of the upper and lower incisors by a caliper while patient's mandible was shifted towards the affected TMJ. Three measurements were performed, and their average is recorded.
Measurement of Lateral Movement of the mandible away from the affected Temporomandibular joint (TMJ) in millimeters | at baseline (t0)
  Lateral Movement of the mandible away from the affected Temporomandibular joint (LA) was measured as the distance between the midlines of the upper and lower incisors by a caliper while patient's mandible was shifted away from the affected TMJ. Three measurements were performed, and their average is recorded.
Measurement of Lateral Movement of the mandible away from the affected Temporomandibular joint (TMJ) in millimeters | at 1st week (t1)
  Lateral Movement of the mandible away from the affected Temporomandibular joint (LA) was measured as the distance between the midlines of the upper and lower incisors by a caliper while patient's mandible was shifted away from the affected TMJ. Three measurements were performed, and their average is recorded.
Measurement of Lateral Movement of the mandible away from the affected Temporomandibular joint (TMJ) in millimeters | at 1st month (t2)
  Lateral Movement of the mandible away from the affected Temporomandibular joint (LA) was measured as the distance between the midlines of the upper and lower incisors by a caliper while patient's mandible was shifted away from the affected TMJ. Three measurements were performed, and their average is recorded.
Measurement of Lateral Movement of the mandible away from the affected Temporomandibular joint (TMJ) in millimeters | at 3rd month (t3)
  Lateral Movement of the mandible away from the affected Temporomandibular joint (LA) was measured as the distance between the midlines of the upper and lower incisors by a caliper while patient's mandible was shifted away from the affected TMJ. Three measurements were performed, and their average is recorded.
Measurement of Lateral Movement of the mandible away from the affected Temporomandibular joint (TMJ) in millimeters | at 6th month (t4)
  Lateral Movement of the mandible away from the affected Temporomandibular joint (LA) was measured as the distance between the midlines of the upper and lower incisors by a caliper while patient's mandible was shifted away from the affected TMJ. Three measurements were performed, and their average is recorded.
Measurement of protrusive movement of the mandible in millimeters | at baseline (t0)
  Protrusive movement of the mandible was measured as the distance in horizontal direction between the incisal edges of upper and lower incisors by a caliper when mandible moves forward.
Measurement of protrusive movement of the mandible in millimeters | at 1st week (t1)
  Protrusive movement of the mandible was measured as the distance in horizontal direction between the incisal edges of upper and lower incisors by a caliper when mandible moves forward.
Measurement of protrusive movement of the mandible in millimeters | at 1st month (t2)
  Protrusive movement of the mandible was measured as the distance in horizontal direction between the incisal edges of upper and lower incisors by a caliper when mandible moves forward.
Measurement of protrusive movement of the mandible in millimeters | at 3rd month (t3)
  Protrusive movement of the mandible was measured as the distance in horizontal direction between the incisal edges of upper and lower incisors by a caliper when mandible moves forward.
Measurement of protrusive movement of the mandible in millimeters | at 6th month (t4)
  Protrusive movement of the mandible was measured as the distance in horizontal direction between the incisal edges of upper and lower incisors by a caliper when mandible moves forward.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih TASKESEN, Study Chair — Erzincan Binali Yildirim University Faculty of Dentistry
Locations (1):
- Erzincan Ağiz Ve Diş Sağlığı Egt Araş Hastanesi, Erzincan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bayramoglu Z, Tozoglu S. Comparison of single- and double-puncture arthrocentesis for the treatment of temporomandibular joint disorders: A six-month, prospective study. Cranio. 2021 Mar;39(2):151-156. doi: 10.1080/08869634.2019.1603796. Epub 2019 Apr 25. PMID 31021311
- [Result] Senturk MF, Yazici T, Findik Y, Baykul T. Intraoperative comparison of single- and double-puncture techniques in temporomandibular joint arthrocentesis. Int J Oral Maxillofac Surg. 2018 Aug;47(8):1060-1064. doi: 10.1016/j.ijom.2018.03.029. Epub 2018 May 1. PMID 29685386

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-20): https://cdn.clinicaltrials.gov/large-docs/59/NCT04367259/Prot_SAP_000.pdf